CLINICAL TRIAL: NCT05946798
Title: Role of NADPH Oxidase in Microvascular Dysfunction Following GDM
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202303158; 1R01HL169201-01 (NIH)
Record Dates: First submitted 2023-06-29; First posted 2023-07-14 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gestational Diabetes; Oxidative Stress; Vascular Endothelial Function
Keywords: gestational diabetes; postpartum; vascular
MeSH Terms: conditions — Diabetes, Gestational | interventions — Acetylcholine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- local lactated Ringer's perfusion (Placebo Comparator): lactated Ringer's is perfused through the microdialysis fiber to serve as the vehicle control
  Interventions: Drug: Acetylcholine; Drug: Insulin aspart
- local apocynin perfusion (Experimental): local apocynin is perfused through the microdialysis fiber to serve as the NADPH oxidase inhibited experimental treatment
  Interventions: Drug: Acetylcholine; Drug: Insulin aspart
- local L-NAME perfusion (Experimental): local L-NAME is perfused through the microdialysis fiber to inhibit nitric oxide synthase
  Interventions: Drug: Acetylcholine; Drug: Insulin aspart
- local apocynin + L-NAME perfusion (Experimental): local apocynin and L-NAME are perfused through the microdialysis fiber for dual inhibition of NADPH oxidase and nitric oxide synthase
  Interventions: Drug: Acetylcholine; Drug: Insulin aspart

INTERVENTIONS:
Drug: Acetylcholine — acetylcholine is perfused at 10 ascending concentrations (10^-10M - 10^-1 M) for 5 minutes each
Drug: Insulin aspart — insulin aspart is perfused at 5 ascending concentrations (10^-8M - 10^-4 M) for 10 minutes each

SUMMARY:
The purpose of this investigation is to examine NADPH oxidase as a source of reactive oxygen species contributing to aberrant microvascular function in otherwise healthy women with a history of GDM.

DETAILED DESCRIPTION:
Women with a history of gestational diabetes mellitus (GDM) are at a 2-fold greater risk for the development of overt cardiovascular disease (CVD) following the effected pregnancy. While subsequent development of type II diabetes elevates this risk, prior GDM is an independent risk factor for CVD morbidity, particularly within the first decade postpartum. GDM is associated with impaired endothelial function during pregnancy and decrements in macro- and microvascular function persist postpartum, despite the remission of insulin resistance following delivery. Collectively, while the association between GDM and elevated lifetime CVD risk is clear, and available evidence demonstrates a link between GDM and vascular dysfunction in the decade following pregnancy, the mechanisms mediating this persistent dysfunction remain unexamined.

The purpose of this investigation is to examine NADPH oxidase as a source of reactive oxygen species contributing to aberrant microvascular function in otherwise healthy women with a history of GDM.

In this study, the investigators use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) they examine the blood vessels in a dime-sized area of the skin in women who have had GDM. As a compliment to these measures, the investigators also collect endothelial cells from an antecubital vein and measure NADPH oxidase expression and markers of oxidative stress in these cells.

ELIGIBILITY:
INCLUSION CRITERIA:

* 18 years or older
* pregnant within 5 years of the study visit
* had gestational diabetes diagnosed by their obstetrician and confirmed according to the American College of Obstetricians and Gynecologists criteria for gestational diabetes.
* or without a history of gestational diabetes

EXCLUSION CRITERIA:

* skin diseases
* current tobacco or electronic cigarette/vape pen use,
* diagnosed or suspected hepatic or metabolic disease including diabetes,
* statin or other cholesterol-lowering medication,
* current antihypertensive medication,
* history of preeclampsia or gestational hypertension,
* current pregnancy,
* body mass index <18.5 kg/m2,
* allergy to materials used during the experiment.(e.g. latex),
* known allergies to study drugs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
microvascular acetylcholine-mediated dilation | at the study visit, an average of 4 hours
  cutaneous vascular vasodilator responses to acetylcholine perfusion in lactated Ringer's, apocynin, L-NAME, and apocynin+L-NAME treated microdialysis sites
microvascular insulin-mediated dilation | at the study visit, an average of 4 hours
  cutaneous vascular vasodilator responses to insulin perfusion in lactated Ringer's, apocynin, L-NAME, and apocynin+L-NAME treated microdialysis sites

SECONDARY OUTCOMES:
endothelial cell NADPH oxidase expression | at the study visit, an average of 4 hours
  NADPH oxidase expression in biopsied endothelial cells

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States